CLINICAL TRIAL: NCT04553055
Title: Assessment of Community Pharmacies Related Antibiotic Misuse and Application of Infection Control Measures During COVID-19 Pandemic
Brief Title: Antibiotic Misuse During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, principle investigator, Beni-Suef University
Other Study IDs: AA86
Record Dates: First submitted 2020-09-15; First posted 2020-09-17 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: coronavirus; observational survey; antibiotics; Egypt
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- community pharmacists
  Interventions: Other: online questionnaires

INTERVENTIONS:
Other: online questionnaires — questionnaire (with detailed questions including how/when/which/for how long antibiotics are prescribed)

SUMMARY:
Evaluating the important role of the community pharmacists in pandemics like covid-19 and to find whether there was a misuse of antibiotics during the pandemic or not and to define the reasons behind this misuse if any present.

DETAILED DESCRIPTION:
Community pharmacy in Egypt is considered as the frontline health care system that is easily and freely accessible by the patients, in this pandemic and due to the current circumstances from closing most general hospitals in front of the public, and with the government applying curfew long hours, community pharmacists were the only healthcare providers available for most patients. Their role will not be restricted to delivering medication but expands to monitoring patient conditions especially those with chronic diseases and patient counseling and education clarifying any misunderstanding concerning covid1-19 medication. The present study includes a questionnaire (with detailed questions including how/when/which/for how long antibiotics are prescribed) that is addressed for community pharmacists who dealt with covid-19 patients during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* All community pharmacists worked during the pandemic and dealt with covid-19 patients inside their pharmacies are welcomed to participate

Exclusion Criteria:

* Clinical and hospital pharmacists- other medical staff- pharmacist assistant

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community pharmacists worked during the pandemic and dealt with covid-19 patients inside their pharmacies are welcomed to participate
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
antibiotic misuse | 15-20 days
  using a questionnaire and direct interviews to evaluate the important role of community pharmacist in pandemics like covid-19 and to assess antibiotic misuse during the pandemic or not and to define the reasons behind this misuse if any present

CONTACTS AND LOCATIONS:
Overall Officials: Hoda M Rabie, PHD, Study Chair — lecturer
Locations (1):
- BeniSuefU, Cairo, BeniSuef, Egypt

IPD SHARING:
Plan to Share IPD: No